CLINICAL TRIAL: NCT01742481
Title: Childhood Cancer Survivor Program to Empower Action in Care
Brief Title: Study to Education Childhood Cancer Survivors About Survivorship Care
Acronym: SPEAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Dr. Lisa Sharp, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K23CA124451 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Cancer
Keywords: childhood cancer survivors; long-term follow-up care; health communication; ethnic/racial minorities; longterm survivors
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and empowerment program (Experimental): Three group sessions delivered once per week over three weeks. Education on late effects of treatment, survivorship care, how to request medical records, and role playing on how to talk to a provider about childhood cancer health risks
  Interventions: Behavioral: Education and empowerment
- self-guided empowerment and education (Placebo Comparator): participants have information packet but receive no individualized support or assistance
  Interventions: Behavioral: Education and empowerment

INTERVENTIONS:
Behavioral: Education and empowerment — Three group sessions delivered once per week over three weeks. Education on late effects of treatment, survivorship care, how to request medical records, and role playing on how to talk to a provider about childhood cancer health risks

SUMMARY:
The proposed study is part of a career development award. The first two phases of research involve collaborating with adult survivors of childhood cancer representing both sexes and three ethnic/racial groups (African American, Hispanic, and White). THe collaboration will focus upon developing educational material that is helpful in teaching survivors about health risks related to cancer treatments and about survivorship care. The third phase is a randomized controlled trial that will randomly (like a flip of coin)place survivors into one of two groups. One group will meet in -person with a group leader three times, once each week over three weeks. The other group will receive an information packet that contains websites, books, and resources similar to content provided in-person within a group format to the other group. The goal is to help adult survivors get involved in specialized healthcare so they can remain healthy. This involves getting a copy of their medical record to understand what treatments they received and working with health providers to get an individualized survivorship care plan.

DETAILED DESCRIPTION:
The proposed study includes three aims: intervention development using focus groups, intervention refinement based upon a pre-pilot, and a randomized controlled pilot study of the final intervention. All participants are adult survivors of childhood cancer, males and females from three ethnic backgrounds (Black, Hispanic, White). The randomized control pilot is designed to assess the acceptibility/feasibility of a community-based intervention to engage childhood cancer survivors more actively in cancer follow-up care. Pilot data on outcome measures will provide data parameters (e.g. means and variances of groups) for accurate power analyses and sample size calculation to support a subsequent efficacy trial.

Relevance: This project is a critical initial step towards addressing systemic problems in transition of care and has the potential to decrease morbidity of adult childhood cancer survivors.

Outcomes include: knowledge of late effects and follow-up care, uncertainty related to 1) relapse, 2) secondary cancers, and 3) late effects, perceived efficacy to communicate with physician, access to childhood medical records, self-efficacy to obtain medical records, and the number of completed health care visits at a six month follow-up interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any childhood cancer excluding CNS prior to age of 18 years
* Completed treatment at least 5 years ago
* Currently cancer free and 18 years or older
* Self-identifies as African American, Hispanic/Latino, or White

Exclusion Criteria:

* Ever seen for risk-based follow-up care as an adult (18 or older)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
scheduling a survivorship visit | 6 months
  Patient report of setting up an appointment at one of the three long-term follow-up clinics in Chicago or setting up an appointment with a physician who is working on a survivorship plan with the patient.

SECONDARY OUTCOMES:
requesting and obtaining medical records from pediatric oncology | 6 months
  Filling out a medical record request form and submitting the form to the pediatric oncology hospital. This may be done by the survivor or the physician.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States